CLINICAL TRIAL: NCT03560414
Title: Study of High - Flux Plasma Diafiltration Based on Plasma - Saved Mode in the Treatment of Patients With Hepatic Failure
Brief Title: The Plasma Diafiltration Therapy of Hepatic Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Principal Investigator, Dongliang Li, professor, Fuzhou General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017L09
Record Dates: First submitted 2018-02-18; First posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Hepatic Failure; Plasma Exchange
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- simple plasma exchange group (Experimental): The mode is CVVH in CRRT machine, the treatment duration is 2h-3h, the application plasma volume is 40ml/Kg, the replacement fluid flow rate is 1000ml/h, the blood flow rate is 100-140 ml/min, and the ultrafiltration volume is 0ml/h.
  Interventions: Procedure: simple plasma exchange
- conventional PDF treatment group (Active Comparator): The mode of conventional PDF treatment group is CVVHDF in CRRT machine, and the duration of treatment is 3 hours. the application plasma volume 1500 ml . The replacement fluid flow rate is 500 ml/h, the dialysate flow rate is 3000 ml/h, the blood flow rate is 100-140 ml/min, and the ultrafiltration volume is 0 ml/h.
  Interventions: Procedure: conventional PDF treatment group
- less plasma PDF treatment group (Active Comparator): The mode of conventional PDF treatment group is also CVVHDF in CRRT machine, and the duration of treatment is 3h. All patients are required to apply plasma 1000ml. Use plasma substitutes: 300ml NS+200ml 5% albumin. The replacement fluid flow rate is 500 ml/h, the dialysate flow rate is 3000 ml/h, the blood flow rate is 100-140 ml/min, and the ultrafiltration volume is 0 ml/h.
  Interventions: Procedure: less plasma PDF treatment group

INTERVENTIONS:
Procedure: simple plasma exchange — simple plasma exchange treatment
  Arms: simple plasma exchange group
Procedure: conventional PDF treatment group — conventional PDF treatment group
  Arms: conventional PDF treatment group
Procedure: less plasma PDF treatment group — less plasma Plasma diafiltration treatment
  Arms: less plasma PDF treatment group

SUMMARY:
At present, there is no comparative study between the simple plasma exchange and plasma diafiltration (PDF), and no further exploration of optimal plasma dose in PDF treatment. Therefore, this prospective randomized cohort study aims to compare the safety and effectiveness of the tree groups（simple plasma exchange group, conventional PDF treatment group, less plasma PDF treatment group）by collecting SOFA score, 3-month survival rate, MELD score, and the times of artificial liver treatment , blood cell variables, cytokines(e.g. TNFα ), pre- and post-treatment plasma ammonia levels. Thus, it is to provide a safer and more effective artificial liver treatment with less plasma dose.

ELIGIBILITY:
Inclusion Criteria:

* hepatic failure on Medium period
* Model for End-Stage Liver Disease (MELD) <30 and >20
* age > 18 years and <70years
* Written informed consent

Exclusion Criteria:

* Active bleeding or disseminated intravascular coagulation
* allergic to blood products or drugs such as plasma, heparin and protamine
* hemodynamic instability
* cardiovascular and cerebrovascular accidental infarction instability Period
* extravascular hemolysis
* severe sepsis
* Tumor on ultrasonography, CT or MRI examination
* Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Model for end-stage liver disease （MELD score） | month 3
  MRLD=R=3.8ln[TBIL(mg/dl)]+11.2ln(INR)+9.6ln [Cr(mg/dl)]+6.4(etiology：Bile or alcoholic 0，others 1)。

SECONDARY OUTCOMES:
cytokine | Month 3
  The concentration of cytokines（TNF-α、IL-６、IL-８、IL-10）will be tested
blood platelet count | Month 3
  To observe the changes in platelet count before and after the treatment
the number of artificial liver treatment | Month3
  Count the number of artificial liver treatments during hospitalization
the concentration of plasma ammonia | Month 3
  To observe the changes of plasma ammonia before and after the treatment
sequential organ failure assessment score（SOFA score） | Month 3
  PaO₂（0：>53.33，1：39-53.33，2：26.66-40，3：13.33-26.67，4：≤13.33）；Platelet count（10/L）（0：>150，1：101-150，2：51-100，3：21-50，4：<21）；Respiratory support（3：NO，4：yes）；TBIL（0：<20，1：20-32，2：33-101，3：102-204，4：>204）；Glasgow Coma Scale（0：15，1：13～14，2：10～12，3：6～9，4：<6）；Cr(umol/L)（0：<110，1：110-170，2：171-299，3：300-440，4：>440）；Level of hypotension (vasopressor status for ≥1 hr)（0：No hypotension；1：MAP <70，2：On vasopressors, dopamine <5 µg/kg/min OR dobutamine (any dose)，3：Dopamine >5 µg/kg/min OR Epi/Norepi <0.1µg/kg/min；4：Dopamine >15 µg/kg/min OR Epi/Norepi >0.1 µg/kg/min）
survival rate | Month 3
  To count the survival rate after the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Fuzhou General Hospital, Xiamen Univ, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No